CLINICAL TRIAL: NCT02772250
Title: Effecacy of Face-to-face Bowel Preparation for Afternoon Colonoscopy: a Randomised Clinical Trial
Brief Title: Bowel Preparation by Face-to-face Re-education on the Day of Colonoscopy for Outpatient: a RCT
Acronym: FFRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, PhD,MD, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016SDU-QILU-04
Record Dates: First submitted 2016-05-07; First posted 2016-05-13 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Bowel Preparation
Keywords: bowel preparation; polyethylene glycol; face-to-face re-education; telephone re-education; Boston Bowel Preparation Scale

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telephone re-education(TRE) (Active Comparator): Subjects who are randomized into this group receive regular instructions at the time of their appointment to discuss colonoscopy (a nurse provides education of 5 minutes and meanwhilet sent a bookle to the patient) and a TRE which was conducted by a investigator at 15:00-17:00 on the day before colonoscopy.
  Interventions: Behavioral: telephone re-education(TRE)
- face-to-face re-education (FFRE) (Experimental): Subjects who are randomized into this group receive regular instructions on the day of their appointment to discuss colonoscopy and also a FFRE which was conducted by a investigator on the same-day of procedure at hospital.
  Interventions: Behavioral: face-to-face re-education (FFRE)

INTERVENTIONS:
Behavioral: telephone re-education(TRE) — Subjects who are randomized into this group receive regular instructions at the time of their appointment to discuss colonoscopy (a nurse provides education of 5 minutes and meanwhilet sent a bookle to the patient) and a TRE which was conducted by one investigator at 15:00-17:00 on the day before colonoscopy.
  Arms: telephone re-education(TRE)
Behavioral: face-to-face re-education (FFRE) — Subjects who are randomized into this group receive regular instructions on the day of their appointment to discuss colonoscopy and also a FFRE which was conducted by a investigator on the same-day of procedure at hospital.
  Arms: face-to-face re-education (FFRE)

SUMMARY:
The study compares the efficacy of bowel preparation between the face-to-face re-education(FFRE group) and normal education (no-FFRE group) in patients.

DETAILED DESCRIPTION:
Despite advances in bowel preparation methods,bowel preparation is inadequate in up to one-third of all colonoscopies in reported series.Inadequate bowel cleansing results in negative consequences for the examination, including incomplete visualisation of the colon, missed lesions, procedural difficulties, prolonged procedure time and reduced time interval until follow-up, and an estimated 12-22% increase in overall colonoscopy cost.

The adequacy of a bowel preparation is closely linked to patient compliance with both dietary and purge instructions.One study performed in Asia showed that non-compliance with bowel preparation instructions, lower education level, and a long wait for the colonoscopy appointment were independent risk factors for poor bowel preparation. Another study performed in China showed that telephone re-education（TRE) about the details of bowel preparation on the day before colonoscopy significantly improved the quality of bowel preparation and PDR. So,it is reasonable to hypothesise that efforts to improve education and maximise patient compliance during the preparatory period will enhance the efficacy of bowel preparation.

The study compares the efficacy of bowel preparation between the face-to-face re-education (FFRE group) and telephone re-education (TRE group) in patients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 18-80 years undergoing colonoscopy who had provided written informed consent

Exclusion Criteria:

* history of colorectal surgery
* severe colonic stricture or obstructing tumour
* dysphagia
* compromised swallowing reflex or mental status
* significant gastroparesis or gastric outlet obstruction or ileus
* known or suspected bowel obstruction or perforation
* severe chronic renal failure (creatinine clearance<30 ml/min)
* severe congestive heart failure (New York Heart Association class III or IV)
* uncontrolled hypertension (systolic blood pressure>170 mm Hg, diastolic blood pressure>100 mm Hg)
* toxic colitis or megacolon
* dehydration
* disturbance of electrolytes
* pregnancy or lactation
* unable to give informed consent
* haemodynamically unstable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation quality at the time of colonoscopy defined by Boston Bowel Preparation Scale rating scores≥6 among 2 groups. | 5 months
  This is an established rating scale to evaluate the quality of bowel prep. The ratings will be compared among the 2 groups.

SECONDARY OUTCOMES:
Rate of compliance with instructions among 2 groups | 5 months
  Compliance was scored on a 3-grade scale based on the intake of bowel solution: 0 = optimal (intake of 100% of the solution); 1 = good (intake of ≥75% of the solution); 2 = poor (intake of <75% of the solution).

OTHER OUTCOMES:
Willingness to repeat bowel preparation among 2 groups. | 5 months
  The willingness to repeat the same bowel preparation,a patient's subjective evaluation of the bowel preparation was recorded by a questionnaire
Polyp detection rate among 2 groups. | 5 months
  Polyp detection rate was defined as the proportion of patients with at least one polyp.
Withdrawal time among 2 groups. | 5 months
  Withdrawal time from ileocecum, not including the time of treatment and biopsy for polyps.
Caecal intubation rate among 2 groups. | 5 months
  Caecal intubation rate is defined the proportion of patients with caecal intubation.

CONTACTS AND LOCATIONS:
Overall Officials: li yanqing, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China